CLINICAL TRIAL: NCT04221178
Title: A Single-Arm, Prospective Study of Maintenance Therapy Cessation for Patients With Multiple Myeloma in Sustained MRD-Negative Remissions
Brief Title: Stopping Maintenance Therapy in People With Multiple Myeloma in MRD-Negative Remission
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-422
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Plasma Cell Myeloma
Keywords: Plasma Cell Myeloma; MRD-Negative; MRD-Negative Remission; Memorial Sloan Kettering Cancer Center; 19-422
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRD-Negative Participants
  Interventions: Other: Cessation of continuous matinenace therapy

INTERVENTIONS:
Other: Cessation of continuous matinenace therapy — Cessation of maintenance therapy for participants in sustained MRD-negative remission while under careful observation

SUMMARY:
This study will test whether stopping maintenance therapy in people with multiple myeloma in MRD-negative remission has the same effect on disease control as continuing this therapy. The study will look at whether people currently on maintenance therapy can safely stop this treatment and continue with active surveillance instead while keeping their MRD-negative remission status for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plasma cell myeloma treated with any number of prior lines of therapy, who at the time of study enrollment have had sustained MRD-negativity at a given timepoint and a subsequent time point with an interval of 3 or more years while on continuous maintenance therapy. MRD-negativity is defined per the International Myeloma Working Group Consensus Panel.
* MRD positivity will be defined by detection of 1 or more neoplastic plasma cells in 10^5 nucleated cells by flow cytometry as per IMWG criteria (i.e., sensitivity of 10-5)
* Age >/= 18 years with ECOG performance status </= 2
* Patients must be able to understand and be willing to sign a voluntary informed consent form and agree to compliance with the protocol schedule; with the knowledge that they may withdraw consent at any time without impact on future medical care

Exclusion Criteria:

* Patients found to be MRD-positive at time of screening
* Patients with plasma cell leukemia or other disorder of plasma cell neoplasm
* Patient who are receiving other therapy with the intent of treating myeloma with the exception of bisphosphonates
* Patients being treated for another, potentially life-limiting malignancy with 3-year lead-in to study enrollment, with the exception of non-melanoma skin cancer or in situ malignancy or malignancies that have received definitive curative therapy
* Prior organ transplant or condition requiring immunosuppressive therapy
* Prior allogeneic hematopoietic cell transplant
* Patients with any other ongoing, concomitant, comorbid illness including but not limited to uncontrolled diabetes, NYHA class III or IV heart failure, uncontrolled coronary artery disease/arrhythmia, psychiatric or social disorder that would compromise compliance with the study schema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted at MSKCC. Efforts will be made to ensure that women and minority groups are adequately represented in this trial. All patients will be seen by MSKCC myeloma physicians and associated MSKCC co-investigators, enrolled and registered at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Maintaining a MRD-negative state for one year of enrolling on this study

CONTACTS AND LOCATIONS:
Overall Officials: Neha Korde, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org